CLINICAL TRIAL: NCT04478214
Title: The Strategic Use of Hyaluronic Acid Fillers and Neurotoxin to Influence Gender Perception in Transgender Individuals
Status: Completed | Type: Observational
Sponsor: Mountain Dermatology Specialists (Other)
Responsible Party: Principal Investigator, Lauren Bonati, Principle Investigator, Mountain Dermatology Specialists
Other Study IDs: MountainDermatology
Record Dates: First submitted 2019-08-16; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Gender Dysphoria
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational survey study of transgender individuals who have undergone cosmetic neurotoxin and soft tissue filler for the purpose of influencing gender perception.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female transgender volunteer
* Has the desire to alter gender perception and is seeking treatment with neurotoxin and soft tissue filler
* Subjects with an already existing treatment plan
* Willing to sign photography release, with the understanding the de-identified photographs may be used in medical publications or presentations for the purposes of education
* Females of childbearing potential who are sexually active are using a reliable method of contraception1 at least one month before the beginning of the study, and throughout the study
* Must be informed about the study objectives and procedures, and be able to understand them
* Willing and able to fulfill the study requirements and schedule
* Willing to give their written informed consent

Exclusion Criteria:

* Individuals who underwent a neurotoxin procedure on the face within 6 months of study start
* Individuals who underwent an injectable filler procedure on the face within 1 year of study start
* Individuals who underwent surgical procedure on the face for the purpose of gender reassignment or cosmetic enhancement at any point in time before study start Individuals who have planned cosmetic treatments or surgeries during the course of the study
* Individuals with dental procedures performed 30 days before, during, or 30 days after the course of the study
* Individuals who participated within the 30 days before inclusion or currently participating in another clinical study involving the investigational areas
* Individuals with known or suspected defect of healing
* Individuals with any disease state or inappropriate physical skin condition that might impair evaluations or increase the health risk to the subject by participation in the opinion of the Investigator
* Individuals unable to be contacted by phone in case of emergency
* Individuals who are currently participating in any other clinical trial or have participated in any clinical trial involving the investigation area within 30 days prior to inclusion into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2 healthy transgender volunteers age 18-65, of any skin type, with the desire to alter gender perception, and are already scheduled for standard of care treatments will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Self perceived gender perception | 4 weeks
  subject reported gender perception on a novel Self-perceived gender perception scale, before and after previously conducted cosmetic treatments. The scale exists on a spectrum of 100% male to 100% female in appearance. Pt will rate themselves along this scale in accordance with their physical appearance as it relates to self-perceived gender.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Bonati, MD, Principal Investigator — Skin Care Physicians
Locations (1):
- Skin Care Physicians, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided